CLINICAL TRIAL: NCT04546594
Title: Collection of Epidemiological Data on Pain Related to Orthopedic, Thoracic or Gynecological Surgery
Brief Title: Epidemiological Data on Pain
Acronym: ALGOBASES
Status: Withdrawn | Type: Observational
Why Stopped: LACK OF RESOURCES
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: RNI_2018_76; 2020-A01112-37 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-09

CONDITIONS: Orthopedic Disorder; Thoracic; Gynecological; Surgery (Previous), Causing Obstructed Labor, Affecting Fetus; Pain
Keywords: Pain,; perioperative pain; epidemiology; predictive factors
MeSH Terms: conditions — Musculoskeletal Diseases; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Orthopedic surgery
- Thoracic surgery
- Gynecological surgery

SUMMARY:
The ALGOBASES project is an observational epidemiological study of pain through the collection of pain evaluation questionnaires and information with the aim of creating a descriptive "pain" evaluation in all patients who need to benefit from orthopedic, thoracic or gynecological surgery. The painful symptomatology will thus be evaluated in all its dimensions (demographic data, physical, psychological, socio-cultural components) and linked to the pathology justifying the specialized care. It is planned to collect the same data at each subsequent event in order to allow the determination of predictive factors, pain trajectories according to the type of surgery, and the profile of subjects at risk of acute or chronic postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 17 years old Patient needing orthopedic surgery Patient needing gynecological surgery Patient needing thoracic surgery Patient who has given written consent to participate in the trial. Socially insured patient Patient willing to comply with all study procedures and study duration

Exclusion Criteria:

* Age under 18 years old
* Non-communicating patient
* Patient does not understand French
* Patient without social protection
* Patient refusing to participate

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients consulting at the university hospital of Lille and needing orthopedic, thoracic, gynecological surgical management with or without painful symptoms and chronic painful patients in the context of organ pathologies.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Descriptive analysis of the typology of pain in patients needing surgery. | Baseline
  The typology of pain will be analyzed on the basis of responses to questionnaires on the affective and sensory dimension of pain, quality of life, depression, anxiety and catastrophizing

SECONDARY OUTCOMES:
Descriptive analysis of specific symptomatology of pain Description of the general and painful symptomatology in patients needing surgery. | follow-up over a period of five years during post-operative or pain medical consultation
  Describe the specific symptomatology of pain separately according to the 3 pathologies: patients needing orthopedic, thoracic and gynecological surgery.
Pain Catastrophizing Scale (PCS) according to pain | Baseline and follow-up over a period of five years during post-operative or pain medical consultation
Hospital Anxiety Depression scale (HAD) according to pain | Baseline and follow-up over a period of five years during post-operative or pain medical consultation
EQD5 according to pain | Baseline and follow-up over a period of five years during post-operative or pain medical consultation
Identification of factors predictive of acute or chronic pain. | Baseline and at three months, six months, one year
  The presence of pain will be defined by the presence of severe pain and/or the presence of neuropathic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Wattier, MD, Principal Investigator — University Hospital, Lille